CLINICAL TRIAL: NCT01342588
Title: Accuracy of Lumbar Pedicle Screw Placement Assisted With Continuous Pulse-train Stimulation During Track Creation and Screw Insertion
Brief Title: Accuracy of Lumbar Pedicle Screw Placement Assisted With Continuous Pulse-train Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Galvan Hernandez Ernesto Eduardo, Organizational affiliation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABC-11-03
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Spine Pedicle Screw Placement
Keywords: Pedicle screws; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical stimulation (Experimental): Only arm of the study, the experimental
  Interventions: Procedure: Electric pulse train stimulation

INTERVENTIONS:
Procedure: Electric pulse train stimulation — Electric pulse train stimulation of regular probes and screw drivers used in track creation and screw placement Using a standard neurophysiological work station, a series of square wave pulses will be delivered through standard probes and screw drivers using an alligator clip during pedicle probing and screw insertion (4 Hz for 50-200 μsec at 10-30 μAmp)

SUMMARY:
The purpose of this study is to establish the accuracy of pedicle positioning using continuous electrical pulse during screwing. Additionally, the investigators evaluate if this maneuver can prevent neurological injury during track creation and screwing in lumbar and thoracic spine instrumentation surgery

DETAILED DESCRIPTION:
Pedicle screw instrumentation as part of spine surgery is a recurrent technique used for most of spine surgeons. Since its description by Boucher in 1959 and its popularization later by Roy-Camille, has been considered a technique that demands great anatomy knowledge and some grade of expertise. Even in experienced hands the misplacement of pedicle screws could have an incidence of 10-40% (average of 20%). Medially misplacements during track creation and screw insertion are the most feared complications, because the anatomic relationship between medial pedicle wall and neural structures. The first attempt to use continuous electrical stimulation during pedicle track creation and screw insertion was communicated in 1997 by Welch WC, et al. In that study they used the bone impedance as a direct measurement of pedicle wall integrity; unfortunately they used inhaled anesthetics and assessed the final screw position with plain X-rays. They reported a sensibility and specificity of 98% and 99% respectively. The great limitation for this study is its assessment of screw accuracy performed by plain X-rays, now a days the best way to do it is with computed tomography (CT).

After the Welch report, a couple of studies more have used similar techniques in the thoracic spine trying to avoid neurological injuries during pedicle screw insertion, but none described the use of continuous train pulses during screwing.

The present study pretends to evaluate the final accuracy and trans-operative usefulness of the pulse train stimulation during track creation and screw insertion using intra venous anesthetic agents and CT scans to assess the integrity of pedicle walls

ELIGIBILITY:
Inclusion Criteria:

* Any patient who needs pedicle screw placement for any spine condition

Exclusion Criteria:

* Previous spine surgery
* Pedicle fracture documented before or during surgery.
* Preoperative identified neurological deficit of the nerve roots close to the instrumented levels

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Intra operative neurophysiological monitoring (IONM) alert | Participants will be followed for the duration of surgical procedure, an expected average of 3-4 hours
  - Continuous electrical stimulation delivered by a wire connected to the surgical instruments only during pedicle track creation and screw placement combined with neurophysiological monitoring will let us identify any IONM alert, defined as nerve irritation or a decrease in voltage and/or amplitude response. This is a single and immediate measurement obtained at surgery during spinal screw placement.

SECONDARY OUTCOMES:
Pedicle screw accuracy | On day 2 after surgery before patient discharge, a CT scan will be performed
  On day 2 post surgery, a CT scan with sagittal, coronal and axial reconstructions will be obtained . The same day of the study, two independent observers will assess the accuracy of screws inside lumbar pedicles, recording in millimeters, any pedicle wall violation on sagittal, axial and coronal views for each screw placed. In that way we could have the accuracy of pedicle screws placed with the proposed technique, before patient discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto E Galvan Hernandez, MD, MsC, Principal Investigator — American British Cowdray Medical Center, Neurological Center
Locations (1):
- American British Cowdray Medical Center, Mexico City, Mexico DF, Mexico

REFERENCES:
- [Background] Roy-Camille R, Saillant G, Mazel C. Internal fixation of the lumbar spine with pedicle screw plating. Clin Orthop Relat Res. 1986 Feb;(203):7-17. PMID 3955999
- [Background] Donohue ML, Murtagh-Schaffer C, Basta J, Moquin RR, Bashir A, Calancie B. Pulse-train stimulation for detecting medial malpositioning of thoracic pedicle screws. Spine (Phila Pa 1976). 2008 May 20;33(12):E378-85. doi: 10.1097/BRS.0b013e31817343c1. PMID 18496333
- [Background] Welch WC, Rose RD, Balzer JR, Jacobs GB. Evaluation with evoked and spontaneous electromyography during lumbar instrumentation: a prospective study. J Neurosurg. 1997 Sep;87(3):397-402. doi: 10.3171/jns.1997.87.3.0397. PMID 9285605
- [Background] Collado-Corona MA, de Leo-Vargas R, Sandoval-Sanchez V, Diaz-Hernandez A, Gutierrez-Sougarret BJ, Shkurovich-Bialik P. Neurophysiological monitoring in spinal cord surgery. Cir Cir. 2009 Sep-Oct;77(5):385-90. PMID 19944028